CLINICAL TRIAL: NCT02494570
Title: A Phase 2 Multi-center Investigation of Efficacy of ABI-009 (Nab-sirolimus) in Patients With Advanced Malignant Perivascular Epithelioid Cell Tumors (PEComa)
Brief Title: A Phase 2 Study of Nab-sirolimus (ABI-009) in Patients With Advanced Malignant PEComa
Acronym: AMPECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEC-001; FD005749 (Other Grant/Funding Number: FDA-OOPD); AMPECT (Other: Aadi)
Expanded Access: NCT03817515 (Approved for marketing)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Malignant PEComa
Keywords: malignant PEComa, perivascular epithelioid cell tumors
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nab-Sirolimus (Experimental): Patients with malignant PEComa received nab-sirolimus on Days 1 and 8 of every 21-day cycle, as a 30-minute IV infusion.
  Interventions: Drug: nab-Sirolimus

INTERVENTIONS:
Drug: nab-Sirolimus — Patients received nab-sirolimus at 100 mg/m2 on Days 1 and 8 of a 21-day cycle by intravenous infusion over 30 minutes.
  Other Names: ABI-009; Fyarro; nab-rapamycin

SUMMARY:
A phase 2 multi-center investigation of efficacy of nab-sirolimus (formerly known as ABI-009 or nab-rapamycin) in patients with advanced malignant perivascular epithelioid cell tumor (PEComa).

DETAILED DESCRIPTION:
This was a phase 2, single-arm, open-label, multi-center study to determine the efficacy and safety profile of nab-sirolimus in patients with advanced malignant PEComa. Patients were required to have measurable disease at baseline (per RECIST v1.1). Eligible patients received nab-sirolimus at 100 mg/m2 by IV infusion (over 30 minutes) weekly for 2 weeks followed by a week of rest (ie, on Day 1 and Day 8 in 21-day cycles). Patients remained on treatment until they experienced progressive disease or unacceptable toxicity, withdrew consent, or physician's decision. Patients who discontinued treatment entered the on-study Follow-up period for survival.

Computed tomography or magnetic resonance imaging (MRI) scans were performed at screening, every 6 weeks for the first year, then every 12 weeks thereafter until the end of treatment. Throughout treatment with nab-sirolimus, patients were routinely assessed for toxicities, the need for dose modifications, and response assessments.

The sample size was targeted to be ~30 patients in order to provide a reasonably precise estimate of the true ORR. Assuming an observed ORR of 30% and a sample size of 30, the lower bound of the 95% confidence interval (CI) for the estimated ORR would exclude values less than 14.7%.

The primary analysis was predefined to be conducted when all patients have had the opportunity to be treated for at least 6 months. The study remained open for 3 additional years and the final analysis occured at study closure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed diagnosis of malignant PEComa that is either metastatic or locally advanced and for which surgery is not a recommended option.
2. Patients must have available tumor block along with the corresponding pathology report (or approximately 30 unstained slides, with a minimum of 16 slides), and/or fresh biopsy to allow retrospective centralized confirmation of malignant PEComa and for mTOR pathway analysis and biomarker analysis.
3. Patients must have one or more measurable target lesions by CT scan or MRI. Measurable disease by RECIST v1.1.
4. Patients must not have been previously treated with an mTOR inhibitor.
5. Prior treatment (investigational or other), chemotherapy, radiotherapy, surgery, or other therapeutic agents (except mTOR inhibitors) is allowed, if completed after 5 half-lives or ≥28 days prior to enrollment, whichever is shorter.
6. Eligible patients, 18 years or older, with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Patients must have the following blood chemistry levels at screening (obtained

   ≤14 days prior to enrollment (local laboratory):
   1. total bilirubin ≤1.5 x upper limit of normal (ULN) mg/dl
   2. AST ≤2.5 x ULN (≤5 x ULN if attributable to liver metastases)
   3. serum creatinine ≤1.5 x ULN
8. Adequate biological parameters as demonstrated by the following blood counts at screening (obtained ≤14 days prior to enrollment, local laboratory):

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L;
   2. Platelet count ≥100,000/mm3 (100 × 109/L);
   3. Hemoglobin ≥9 g/dL.
9. Serum triglyceride <300 mg/dL; serum cholesterol < 350 mg/dL.
10. Male or non-pregnant and non-breast feeding female:

    * Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting IP and while on study medication and have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment.
    * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, even if he has undergone a successful vasectomy.
11. Life expectancy of >3 months, as determined by the investigator.
12. Ability to understand and sign informed consent.
13. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Patients with lymphangioleiomyomatosis (LAM) are excluded.
2. Known active uncontrolled or symptomatic central nervous system (CNS) metastases. A patient with controlled and asymptomatic CNS metastases may participate in this study. As such, the patient must have completed any prior treatment for CNS metastases ≥28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
3. Active gastrointestinal bleeding, if transfusion dependent.
4. Pre-existing thyroid abnormality is allowed provided thyroid function can be controlled with medication.
5. Uncontrolled serious medical or psychiatric illness. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason Score ≤ 6 and postoperative PSA <0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥1 year).
6. Liver-directed therapy within 2 months of enrollment. Prior treatment with radiotherapy (including radio-labeled spheres and/or cyberknife, hepatic arterial embolization (with or without chemotherapy) or cyrotherapy/ablation) is allowed if these therapies did not affect the areas of measurable disease being used for this protocol.
7. Recent infection requiring systemic anti-infective treatment that was completed

   ≤14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
8. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy.
9. Unstable coronary artery disease or myocardial infarction during preceding 6 months.
10. Receiving any concomitant antitumor therapy.
11. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
12. The use of certain medications and illicit drugs within 5 half-lives or 28 days, whichever is shorter prior to the first dose of study drug and for the duration of the study will not be allowed.
13. Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanide) within the 14 days prior to receiving the first dose of ABI-009.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10; Primary Completion 2021-11 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willis Navarro, MD, Study Director — Aadi Bioscience
Locations (9):
- United States (9):
  - Stanford University Medical Center, Palo Alto, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Wagner AJ, Ravi V, Riedel RF, Ganjoo K, Van Tine BA, Chugh R, Cranmer L, Gordon EM, Hornick JL, Du H, Polson KM, Yalamanchili S, DeBoer C, Ding L, Schmid AN, Navarro WH, Kwiatkowski DJ, Dickson MA. A plain language summary of the AMPECT study: nab-sirolimus for advanced malignant perivascular epithelioid cell tumors. Future Oncol. 2026 Jan;22(1):1-13. doi: 10.1080/14796694.2025.2574811. Epub 2025 Dec 22. PMID 41424265
- [Derived] Wagner AJ, Ravi V, Riedel RF, Ganjoo K, Van Tine BA, Chugh R, Cranmer L, Gordon EM, Hornick JL, Du H, Ding L, Schmid AN, Navarro WH, Kwiatkowski DJ, Dickson MA. Phase II Trial of nab-Sirolimus in Patients With Advanced Malignant Perivascular Epithelioid Cell Tumors (AMPECT): Long-Term Efficacy and Safety Update. J Clin Oncol. 2024 May 1;42(13):1472-1476. doi: 10.1200/JCO.23.02266. Epub 2024 Mar 1. PMID 38427923
- [Derived] Wagner AJ, Ravi V, Riedel RF, Ganjoo K, Van Tine BA, Chugh R, Cranmer L, Gordon EM, Hornick JL, Du H, Grigorian B, Schmid AN, Hou S, Harris K, Kwiatkowski DJ, Desai NP, Dickson MA. nab-Sirolimus for Patients With Malignant Perivascular Epithelioid Cell Tumors. J Clin Oncol. 2021 Nov 20;39(33):3660-3670. doi: 10.1200/JCO.21.01728. Epub 2021 Oct 12. PMID 34637337

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Nab-Sirolimus: Patients with malignant PEComa were treated with 100 mg/m2 nab-sirolimus (30 mins IV infusion) on Days 1 and 8 in a 21-day cycle.
Period: Overall Study
Arm/Group | Experimental: Nab-Sirolimus
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: patients treated with nab-sirolimus (N = 34)
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 60 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
ECOG Performance Score [Count of Participants; unit: Participants]
  0 (Fully active, able to carry on all pre-disease performance without restriction) | 26
  1 (Restricted in physically strenuous activity but ambulatory and able to carry out light work) | 8
Metastatic PEComa [Count of Participants; unit: Participants] — For the assessment of overall tumor burden and measurable advanced disease (metastatic or locally advanced) at baseline, computed tomography (CT) or contrast enhanced magnetic resonance imaging (MRI) could be used, as long as the same modality was used throughout the study. Baseline scans were done at done within 4 weeks of starting therapy and must have included (as clinically indicated), chest, abdominal, and pelvic CT or MRI.
  Participants | 29
Locally Advanced, Inoperable PEComa [Count of Participants; unit: Participants] — For the assessment of overall tumor burden and measurable advanced disease (metastatic or locally advanced) at baseline, computed tomography (CT) or contrast enhanced magnetic resonance imaging (MRI) could be used, as long as the same modality was used throughout the study. Baseline scans were done at done within 4 weeks of starting therapy and must have included (as clinically indicated), chest, abdominal, and pelvic CT or MRI.
  Participants | 5
Prior Systemic Therapy for Advanced PEComa [Count of Participants; unit: Participants] | 4
Primary Tumor Location of PEComa [Count of Participants; unit: Participants] — PEComa can be located at various anatomic sites.
  Participants
    Uterus | 8
    Pelvis, extrauterine | 6
    Retroperitoneum | 6
    Lung | 4
    Kidney | 4
    Aorta | 1
    Brain | 1
    Liver | 1
    Muscle | 1
    Ovary | 1
    Small Bowel | 1
Number of Metastatic Sites [Count of Participants; unit: Participants] — Population: Patients with metastatic lesions n = 29.
  Participants
    number analyzed (Participants) | 29
    1 metastatic site (best) | 11
    2 metastatic sites | 9
    3 metastatic sites | 7
    >3 metastatic sites (worst) | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Overall Response Rate (ORR)
Description: Best ORR was assessed by Independent Radiology Review using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria. Best overall response was the best response recorded from the start of the study treatment until the end of treatment taking into account the requirement for confirmation.
  Per RECIST v1.1, best overall response assignment depended on the findings of both target and non-target disease and also took into consideration the appearance of new lesions. Overall response rate was defined as the percentage of patients who achieve a confirmed PR or CR per RECIST 1.1. At each timepoint, objective tumor response for target lesions were assessed as such: Complete Response (CR), disappearance of all target lesions, and pathological lymph nodes must have a reduction <10 mm; Partial Response (PR), ≥30% decrease in the sum of the longest diameter of target lesions.
Time Frame: through study completion (up to 72 months)
Population: Efficacy Evaluable Patient Population
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Sirolimus: Patients with malignant PEComa were treated with 100 mg/m2 nab-sirolimus (30 mins IV infusion) on Days 1 and 8 in a 21-day cycle.
Arm/Group | Nab-Sirolimus
Number analyzed (Participants) | 31
Participants
  Best Overall Confirmed Complete Response | 2
  Best Overall Confirmed Partial Response | 10
  Best Overall Stable Disease | 16
  Best Overall Progressive Disease | 3

2. Secondary Outcome: Duration of Response
Description: The time from the start of CR or PR to the first date of documented PD or death.
Time Frame: From Initial response until tumor progression, through study completion (up to 72 months)
Population: Patients with a confirmed partial or complete response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 12
months | 39.7 [6.5 to NA] — Upper limit was not reached due to insufficient number of participants with events

3. Secondary Outcome: Progression-free Survival Rate at 6 Months
Description: The time from the first dose date to the first observation of a disease progression or death due to any cause by 6 mo. Disease progression was assessed radiologically per RECIST v1.1, and was defined as ≥20% increase in the sum of diameters of target lesions, and absolute increase of ≥5 mm. PFS rate at 6 months was summarized using Kaplan-Meier methods (percentage rounded up to 1 digit decimal).
Time Frame: 6 months
Population: Efficacy Evaluable Patient Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 31
percentage of participants | 69.5 [47.6 to 83.7]

4. Secondary Outcome: Progression-free Survival (Median)
Description: The time from the first dose date to the first observation of a disease progression or death due to any cause.
Time Frame: from start of treatment to first documented disease progression, through study completion (up to 72 months)
Population: Efficacy Evaluable Patient Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 31
months | 10.6 [5.5 to 53.1]

5. Secondary Outcome: Overall Survival
Description: Defined as teh time from first dose date to the date of death due to any cause
Time Frame: From start of treatment to date of death (of any cause), through study completion (up to 72 months)
Population: Treated Patient Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 34
months | 53.1 [22.2 to NA] — Upper limit was not reached due to insufficient number of participants with events

6. Post Hoc Outcome: Disease Control Rate
Description: The percentage of patients who achieve confirmed CR or PR or SD ≥12 weeks following study treatment initiation.
Time Frame: through study completion (up to 72 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Nab-Sirolimus
Number analyzed (Participants) | 31
Participants | 10

ADVERSE EVENTS:
Time Frame: Safety and tolerability were monitored through continuous reporting of treatment-emergent and treatment-related adverse events (AEs) and serious AEs throughout the study, from the time the patient signed informed consent until 28 days after the last dose of study drug, up to 72 months.
Arm/Group | Experimental: Nab-Sirolimus
All-Cause Mortality (participants affected / at risk) | 2/34
Serious Adverse Events (participants affected / at risk) | 16/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Nab-Sirolimus (N=34)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pyrexia (Blood and lymphatic system disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Nab-Sirolimus (N=34)
Stomatitis (Gastrointestinal disorders) | 28 (69)
Nausea (Gastrointestinal disorders) | 17 (40)
Diarrhoea (Gastrointestinal disorders) | 16 (39)
Abdominal Pain (Gastrointestinal disorders) | 15 (33)
Vomiting (Gastrointestinal disorders) | 13 (31)
Fatigue (General disorders) | 25 (47)
Edema (General disorders) | 19 (32)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (45)
Decreased appetite (Metabolism and nutrition disorders) | 15 (21)
Hypokalemia (Metabolism and nutrition disorders) | 15 (33)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13 (25)
Hypercholesterolemia (Metabolism and nutrition disorders) | 12 (21)
Anemia (Blood and lymphatic system disorders) | 21 (110)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (37)
Hemorrhage (Blood and lymphatic system disorders) | 11 (28)
Infections (Infections and infestations) | 20 (86)
Taste Disorder (Nervous system disorders) | 12 (25)
Headache (Nervous system disorders) | 12 (24)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (21)
Weight Decreased (Investigations) | 17 (45)
Rash (Skin and subcutaneous tissue disorders) | 23 (55)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (18)
ALT (Investigations) | 9 (20)
AST (Investigations) | 9 (18)
Leukopenia (Blood and lymphatic system disorders) | 9 (43)
Peripheral neuropathy (Nervous system disorders) | 8 (8)
Dizziness (Nervous system disorders) | 7 (11)
Non-infectious pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (22)
Pain (General disorders) | 7 (10)
Lymphopenia (Blood and lymphatic system disorders) | 6 (21)
Dehydration (Metabolism and nutrition disorders) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Neutropenia (Blood and lymphatic system disorders) | 5 (14)
Fracture (General disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (5)
Dental pain (General disorders) | 3 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (4)
Ear pain (Ear and labyrinth disorders) | 2 (4)
Constipation (Musculoskeletal and connective tissue disorders) | 8 (11)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Lipase increased (Investigations) | 10 (20)
Amylase increased (Investigations) | 9 (40)
Creatinine increased (Investigations) | 9 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (11)
Dysgeusia (Nervous system disorders) | 11 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT02494570/Prot_SAP_000.pdf